CLINICAL TRIAL: NCT07068828
Title: The Effect of Mobilization Incentive Protocol Applied to Bariatric Surgery Patients on Physical Mobility, Recovery Quality and Complications
Brief Title: The Effect of Encouraging Patients Undergoing Obesity Surgery to Move on Physical Mobility, Recovery and Negative Effects of Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Yunus Gökkaya, Nurse, MSc, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ERU-SBF-YG-01; BAP-14157 (Other Grant/Funding Number: Erciyes University Scientific Research Projects Unit)
Record Dates: First submitted 2025-07-04; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Physical Activity; Bariatric Surgery; Quality of Recovery; Mobilization
Keywords: bariatric surgery; physical activity; quality of recovery; mobilization
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobilization Encouragement Group (Experimental): Participants in this group receive a mobilization encouragement protocol consisting of a video-based education session before surgery, visual reminders (posters) in their rooms on post-op day 1, and SMS reminders sent to their phones on post-op days 1 and 3. Participants will wear a smart watch starting 8 hours after surgery to track physical activity (step count). The goal is to increase early mobilization, improve recovery quality, and reduce postoperative complications.
  Interventions: Behavioral: Mobilization Encouragement Protocol; Behavioral: Smart Watch for Physical Activity Monitoring
- Standard Care Control Group (Active Comparator): Participants in this group receive routine postoperative care without additional mobilization encouragement. They will also wear a smart watch to monitor physical activity, but will not receive educational videos, posters, or SMS reminders. This group serves as a comparison to evaluate the effect of the mobilization protocol.
  Interventions: Behavioral: Smart Watch for Physical Activity Monitoring

INTERVENTIONS:
Behavioral: Mobilization Encouragement Protocol — This intervention includes a video-based education session delivered before surgery to encourage early mobilization, visual poster reminders in patient rooms on postoperative day 1, and SMS text message reminders sent to patients' phones on postoperative days 1 and 3. Participants will also wear a smart watch starting 8 hours after surgery through postoperative day 3 to monitor physical activity (step count). The goal is to increase physical activity levels, improve recovery quality, and reduce postoperative complications after bariatric surgery.
  Other Names: Postoperative Mobilization Program
  Arms: Mobilization Encouragement Group
Behavioral: Smart Watch for Physical Activity Monitoring — Participants in the control group receive standard postoperative care without additional mobilization encouragement. They wear a smart watch starting 8 hours after surgery through postoperative day 3 to monitor physical activity (step count). However, they do not receive video education, posters, or SMS reminders.
  Other Names: Postoperative Mobilization Program

SUMMARY:
Early mobilization and physical mobility have a critical role in minimizing complications after surgical procedures. Although there are a limited number of studies in the literature on the step count of bariatric surgery patients, there is no study focusing on interventions that promote mobilization in this patient group. The aim of this study was to determine the effect of a mobilization incentive protocol on physical mobility, quality of recovery and complications in patients undergoing bariatric surgery.

This single-blind randomized controlled study will include 70 individuals who underwent bariatric surgery in the General Surgery ward of Kayseri City Hospital between July 2025 and June 2026. Patients will be followed up for 3 days after surgery, starting with the hospitalization process in the clinic before surgery. All participating patients will be administered preoperative patient information form, 6-minute walk test and International Physical Activity Questionnaire. Patients in the intervention group will be shown video-based mobilization training after bariatric surgery. The control group will not receive any intervention. Both groups will wear a smart watch at the time of the first mobilization (8th hour after surgery) and a patient follow-up form will be filled out. A reminder brochure will be hung in their rooms on the 1st postoperative day and a reminder text message will be sent to their cell phones on the 1st and 3rd days. The number of steps will be measured from the smart watch for three days postoperatively, complications will be followed according to the clavien dindo classification system and the Quality of Recovery-15 scale will be applied on the 3rd postoperative day. The analysis of the research data will be performed in IBM SPSS Statistics 26.0 package program. When comparisons between groups are made, parametric tests will be used in the analysis of data showing normal distribution in numerical data, and non-parametric tests will be used in the analysis of data not showing normal distribution. Chi-square test will be used in the analysis of categorical variables.

The lack of protocols to increase mobilization emphasizes the importance and innovativeness of this study. The mobilization promotion protocol is expected to increase the physical activity level (number of steps) of bariatric surgery patients in the postoperative period, improve the quality of recovery and reduce complications. These findings will reveal the importance of mobilization incentive protocol by contributing to postoperative care strategies.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age,
* Can speak and understand Turkish,
* No communication problems,
* Admitted to the clinic for bariatric surgery,
* undergoing elective surgery,
* Who agreed to wear a smartwatch,
* Smartphone users,
* Individuals who volunteered to participate in the study and who do not have physical movement disabilities

Exclusion Criteria:

* In any of the ASA IV and V groups according to the ASA Physical Condition Classification System,
* 6-min walk test contraindicated (unstable angina pectoris within the last month, systolic blood pressure above 180 mmHg, diastolic blood pressure above 100 mmHg, resting heart rate above 120),
* Have any cognitive or neurological impairment that may adversely affect ambulation or cooperation,
* Using a walking aid such as cane, walker, etc. while walking,
* Have a disease that requires assistance with physical movement (e.g. after stroke, limb amputation)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Physical Activity Level (Step Count) | Postoperative 3 days
  Increase in daily step count measured objectively by smart watches in bariatric surgery patients receiving the mobilization encouragement protocol.
  Xiaomi redmi watch 3 active smartwatch is used in the study.The battery lasts 12 days in normal use and 8 days in intensive use. The battery has a capacity of 298 mAh. Bluetooth 5.3 support. It connects to smartphones with Android 6.0 or iOS 12.0 and above versions. After connecting via Bluetooth, the number of steps taken during the day is recorded on the phone. The watch setup requires installing the Mi Fitness (Xiaomi Wear Lite) application and logging in. The application is paired with the QR code on the watch and the watch is connected to the phone via bluetooth.
  Before the patient is mobilized, the patients will be fitted with a smart watch and will be informed about the smart watch and reminded not to take it off. On postoperative day 1, day 2 and day 3, the smartwatch will be checked and the number of steps taken will be recorded

SECONDARY OUTCOMES:
Quality of Recovery | Postoperative day 3
  Improvement in recovery quality assessed by the Quality of Recovery-15 (QoR-15) questionnaire on postoperative day 3.The QoR-15 consists of 15 items in which the patient evaluates pain, physical comfort, physical independence, psychological support and emotional state. Items 11, 12, 13, 14 and 15 are reverse scored. The total score of the unidimensional scale is calculated by summing the scores given for each item. The highest score that can be obtained from the scale is 150 and the lowest score is 0 (zero). A score close to 150 indicates a high quality of recovery
Postoperative Complications | Postoperative 3 days
  Reduction in postoperative complications (e.g., deep vein thrombosis, pulmonary complications, wound healing problems) evaluated using the Clavien-Dindo classification system within 3 days after surgery. In the study, early postoperative complications will be recorded in the Patient Follow-up Chart using the Clavien-Dindo (CD) classification system. According to the CD classification system, postoperative complications are classified into five grades (I-V). In the study, patients will be divided into 2 groups according to CD classification; minor complication group including CD classification grades I to II and major complication group including CD classification grades III to IV.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Yüceler Kaçmaz, Associate Professor Doctor, Study Director — TC Erciyes University

IPD SHARING:
Plan to Share IPD: No
There is no plan